CLINICAL TRIAL: NCT02967848
Title: Liver Function Investigation With Single Photon Emission Computed Tomography After Radiotherapy
Brief Title: Liver Function Investigation With SPECT
Acronym: LiverINSPECT
Status: Active, not recruiting | Type: Observational
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Professor Andrew Kneebone, Associate Professor Andrew Kneebone, Royal North Shore Hospital
Other Study IDs: RESP/16/129
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Liver Cancer, Adult
Keywords: Radiotherapy; Mebrofenin; Liver; Cancer; SPECT
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Cancers in Liver: Adult patients with primary liver cancer or liver metastases from any other histology who will be measured before and after Radiotherapy by '99mTc-mebrofenin hepatobiliary scintigraphy (HBS), Indocyanine Green and Liver Elasticity.
  Interventions: Other: 99mTc-mebrofenin hepatobiliary scintigraphy (HBS); Other: Indocyanine Green; Other: Liver Elasticity

INTERVENTIONS:
Other: 99mTc-mebrofenin hepatobiliary scintigraphy (HBS) — 99mTc-mebrofenin HBS is a SPECT imaging procedure that allows evaluation of global and local liver function. Mebrofenin, bound to albumin, is taken up by hepatocytes in a similar manner to organic anions such as bilirubin. After hepatic uptake, the mebrofenin is excreted into the bile canaliculi. Dynamic imaging tools allow measurement of clearance rates for global function, and 3D SPECT imaging with corresponding CT allows visualisation of the local liver function with respect to anatomy. HBS allows direct visualisation of hepatocyte function.
Other: Indocyanine Green — ICG is a fluorescent dye injected into the patient. The dye is exclusively excreted by the liver. The ICG clearance rate is measured in the finger of the subject.
  Other Names: ICG
Other: Liver Elasticity — This is an Ultrasound measurement of the elasticity of the liver.
  Other Names: Liver FibroScan

SUMMARY:
This is a Phase 1 pilot study to assess feasibility and utility of 99mTc-mebrofenin hepatobiliary scintigraphy for measurement of functional liver change due to radiotherapy.

DETAILED DESCRIPTION:
Patients with cancers of the liver who are not suitable for surgery or chemo/radio embolisation are often treated with stereotactic ablative body radiotherapy (SABR). SABR results in high local control rates but, similar to other treatment modalities, carries risk of damage to healthy surrounding liver. This study aims to use a novel nuclear medicine imaging tracer, 99mTcMebrofenin, to evaluate liver function before and after radiotherapy.

Patients will have a 99mTcMebrofenin scan performed < 2 weeks before radiotherapy and 1 and 6 months after radiotherapy. At the same time points, indocyanine green (ICG) and liver elasticity tests will be performed. These are global measures of liver function, whereas 99mTcMebrofenin is both global and local. From the imaging data, the Investigators will be able to correlate change in local liver function in each sub volume of the liver with the radiotherapy dose it received. The Investigators will be able to thus measure the effect of radiotherapy on global and local liver function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Has provided written Informed Consent for participation in this trial and is willing to comply with the study
* Patients undergoing external beam radiotherapy at Northern Sydney Cancer Centre
* Histologically proven hepatocellular carcinoma or oligometastatic liver metastases (3 or less). Histological diagnosis will be obtained if clinically indicated.
* ECOG performance status 0-2

Exclusion Criteria:

* Previous high-dose radiotherapy to the liver
* Previous SIRT
* Women who are pregnant or lactating
* Unwilling or unable to give informed consent
* No venous access
* Inability to lie supine and still for 30 minutes
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to indocyanine green, including those patients with a history of iodide or seafood allergy (excluded from ICG testing only)
* Pacemaker (excluded from Fibroscan elasticity test only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Liver Cancer patients attending the Northern Sydney Cancer Centre at the Royal North Shore Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-10-19 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in global and local liver function | 3 years
  99mTC-mebrofenin hepatobiliary scintigraphy images after stereotactic ablative body radiotherapy to cancers of the liver. This will be reported as a change in function as a function of delivered radiotherapy dose.

SECONDARY OUTCOMES:
Correlation between 99mTC mebrofenin HBS and various measures of global function | 3 years
  This correlation will be measured using liver elasticity, Indocyanine Green (ICG) and Child-Pugh and Model for End stage Liver Disease (MELD) scores
Relationship between radiological features on CT images and SPECT images | 2 years
  Relationship between radiological features or changes visable on computed tomography (CT) image data and changes in local liver function as observed on 99mTC mebrofenin HBS.
Radiotherapy dose sparing of functional liver | 2 years
  The amount of sparing of dose to functional liver that can be achieved using 99mTC Mebrofenin HBS to guide treatment plan optimisation will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data will be processed remotely at Peter MacCallum Cancer Centre, by the AI, Nicholas Hardcastle.